CLINICAL TRIAL: NCT05994495
Title: Utility, Acceptability and Applicability of a Nucleic Acid Amplification Test (NAAT) in Comparison With Syndromic Approach in the Management of Sexually Transmitted Diseases at Mulago National Referral Hospital in Uganda
Brief Title: Utility and Acceptability of a Molecular Test in the Management of Sexually Transmitted Diseases in Uganda
Acronym: ASTRHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riccardo Serraino (Other)
Collaborators: Societa' Italiana Di Malattie Infettive E Tropicali (Other)
Responsible Party: Sponsor-Investigator, Riccardo Serraino, Fellow, Azienda Ospedaliera Universitaria Mater Domini, Catanzaro
Organization: Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MHREC2023-97
Record Dates: First submitted 2023-08-06; First posted 2023-08-16 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-05

CONDITIONS: Sexually Transmitted Diseases
Keywords: Sexually transmitted diseases; STDs; Low-Middle Income Country; Molecular Test; NUCLEIC ACID AMPLIFICATION TEST; NAAT; Clinical Syndromic Approach; LMIC
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: This is an operational, randomized, open-label trial to assess appropriateness of therapy, diagnostic accuracy, clinical and microbiological outcomes, and acceptability of an etiology approach using a molecular test (NAAT) versus a clinical syndromic approach for the management of STDs in patients followed by a STD clinic of a National Referral Hospital in Kampala, Uganda.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A Molecular test (Experimental): Patients randomized to Arm "A" will be subjected to a microbiological test (either swabs or urine testing by NAAT). After having obtained the result of the molecular test, patients will be prescribed a targeted treatment
  Interventions: Diagnostic Test: nuclear acid amplification tests
- ARM B Clinical Syndromic Approach (Active Comparator): Patients randomized to Arm "B" will be subjected to a molecular test, but they will be treated according to the current guidelines and the best practice using the clinical syndromic approach. So, patients randomized to Arm "B" and their physician also will be blinded to the results of the molecular test
  Interventions: Other: Clinical Syndromic Approach

INTERVENTIONS:
Diagnostic Test: nuclear acid amplification tests — The NAAT test will be performed with Bosch Vivalytic STI test. It is a qualitative Polymerase Chain Reaction-based assay for simultaneous detection of 10 common sexually transmitted pathogens: Herpes simplex virus 1 (HSV 1)- Herpes simplex virus 2 (HSV 2)- Chlamydia trachomatis (CT) - Haemophilus ducreyi (HD)- Mycoplasma genitalium (MG) - Mycoplasma hominis (MH) - Neisseria gonorrhoeae (NG) - Treponema pallidum (TP)- Ureaplasma urealyticum (UU) - Trichomonas vaginalis (TV)
  Other Names: Bosch Vivalytic STI test
  Arms: ARM A Molecular test
Other: Clinical Syndromic Approach — Physical examination
  Arms: ARM B Clinical Syndromic Approach

SUMMARY:
The goal of this clinical trial is to assess utility and acceptability of a molecular test in comparison with clinical syndromic approach in the management of sexually transmitted diseases (STD) at STD clinic of Mulago National Referral Hospital in Uganda.

The main questions it aims to answer are:

* Does new molecular test improve appropriateness of therapy compared with the clinical syndromic approach without or with limited laboratory tests in the management of STDs?
* Are new molecular tests both clinically useful and acceptable in a Low-Middle Income Country for the management of STDs?

Participants will be put into two groups ("A" or "B"):

* Participants in group "A" will have a pus swab collected from urethra or vagina or a urine sample. After the result of the test, patients will be prescribed a specific drug.
* Participants in group "B" will have a pus swab collected from urethra or vagina or a urine sample, but participants in group "B" and their doctor will not know the results of the test. So, participants in group "B" will be given treatment in the standard way, according to the current clinical practice.

DETAILED DESCRIPTION:
Sexually transmitted diseases (STDs) are a major cause of long-term disability. Urethral discharge syndrome (UDS), abnormal vaginal discharge (AVD) and genital ulcer disease (GUD) are very common syndromes in low- and middle-income countries where, due to lack of resources, these syndromes are managed according to a syndromic approach. Appropriate STD diagnosis and treatment are crucial to prevent the transmission and sequelae. No randomized trials have been conducted so far to evaluate clinical usefulness and acceptability of microbiological diagnosis using NAAT in comparison with syndromic approach.

The aims of the study is to evaluate the clinical usefulness of a NAAT in terms of appropriateness of therapy, clinical and microbiological outcomes, diagnostic accuracy, and acceptability in comparison with syndromic approach and to explore whether this test could replace the syndromic approach in the management of STDs at a National Referral Hospital in Uganda. At last, to estimate the actual prevalence of causative agents of STDs in this setting.

In summary final aim is that the results could inform diagnostic guidelines since they may suggest an update of the current recommendations. Investigators speculate that the change in approach would allow a significant improvement in terms of appropriateness of therapy, reduction of the collateral damage, toxicity, and pharmacoeconomics costs.

This is an operational, randomized, open-label trial. Patients will be randomized (using block computerized method) into two Arms ("A" or "B"). Patients randomized to Arm "A" will be subjected to a microbiological test (either swabs or urine testing by NAAT). After having obtained the result of the molecular test, patients will be prescribed a targeted treatment. Patients randomized to Arm "B" will be subjected to a molecular test, but they will be treated according to the current guidelines and the best practice using the clinical syndromic approach. So, patients randomized to Arm "B" and their physician also will be blinded to the results of the molecular test. All the patients randomized to Arm "A" or to Arm "B" will be asked to return after two-three weeks for a control visit. The NAAT test will be performed with Bosch Vivalytic Sexually Transmitted Infection test.

STUDY POPULATION Adults aged 18 years and above presenting with signs and symptoms of STDs at the Mulago Hospital STDs clinic during the study period, who provide written consent to the participation to the study and are diagnosed with UDS, AVD and GUD. Persons belonging to special populations (i.e., female sex workers, MSM) will be analyzed separately.

SAMPLE SIZE Eighty-seven patients (rounded to 90) in each treatment arm are necessary for demonstrating a difference of 0.20 by means of the Fisher's exact test carried out at a significance level of 0.05 (two tailed). The sample size will be increased to 110 patients in each treatment arm for allowing a drop- out rate of about 20%.

SAMPLING METHOD Two groups will be created by a random process and a blinded intervention. The intended sample will be composed by all sequential patients presenting with signs or symptoms suggestive for STDs at the time of screening for inclusion into the trial. Only patients who will satisfy the inclusion and exclusion criteria will be randomized after signing the informed consent. The randomization process will be carried out according to a complete block model. In addition, randomization will be stratified by gender. Any efforts will be put into improving the internal and external validity of the trial.

Data will be collected in an anonymized form: an Identification number will be assigned to each patients. Data will be analyzed by statistical team which will be led by a senior statistician

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females with UDS, AVD and GUD diagnosed as per the current National STD Management Guidelines 201616, who have given informed, written, and signed consent.

Exclusion Criteria:

* All patients presenting with UDS, AVD and GUD who decline informed and written consent.

  * All patients living farther than a 20 km radius from Mulago National Referral Hospital
  * All patients presenting with any syndromes not listed above.
  * Female patients in their menstrual period.
  * Pregnant patients.
  * Patients with a previous infection presenting with recurrence or relapse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Clinical Usefulness | minutes 210
  Proportion of patients with appropriate therapy in each arm. Appropriate therapy will be defined (either as study intervention during consultation in Arm "A" or post-hoc in Arm "B") as the use of a recommended drug or drug combinations which are recommended against the pathogen(s) diagnosed by the molecular test.

SECONDARY OUTCOMES:
Microbiological and clinical cure | weeks 3
  Microbiological cure measured as the percentage of patients who will achieve success at the test of cure performed after two-three weeks from the end of therapy in both arms. For the clinical outcome, we will consider the percentage of patients who will recover from signs and symptoms of the STDs in both arms at the same time-point.
Concordance | Minutes 210
  Percentage of concordant results between the syndromic approach and the NAAT. The diagnosis is considered concordant when at least one pathogen responsible for a specific syndrome (Table 1) diagnosed through the syndromic approach is detected by a molecular testing. The diagnosis is considered not concordant when one or more pathogens responsible for syndromes other than those identified by the syndromic approach, are detected by molecular testing.
Acceptability | Minutes 210
  Percentage of patients who will be sent home the same day with the treatment prescribed according to the molecular test result (Arm "A") or with the treatment according to the syndromic approach (Arm "B"). Patients will not be able to wait for the result of the test and for the targeted therapy will be considered as failure for the primary endpoint. In addition, patients who will drop out from the study will be considered as failure.
  Percentage of patients who will be sent home the same day with the treatment prescribed according to the molecular test result (Arm "A") or with the treatment according to the syndromic approach (Arm "B"). Patients will not be able to wait for the result of the test and for the targeted therapy will be considered as failure for the primary endpoint. In addition, patients who will drop out from the study will be considered as failure.
Prevalence | Months 2
  Prevalence of detected pathogens' genome at the molecular test (overall population).

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Torti, Principal Investigator — Magna Graecia University of Catanzaro, Italy; Patrick Musinguzi, Principal Investigator — Mulago National Referral Hospital, Kampala, Uganda
Locations (1):
- Mulago National Referral Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serraino R, Cesana BM, Morrone HL, Marino GG, Cirillo M, Olivadese V, Kyambadde P, Biriwo LS, Mutebi F, Trecarichi EM, Musinguzi P, Byakika-Kibwika P, Torti C. Utility, acceptability and applicability of a nucleic acid amplification test in comparison with a syndromic approach in the management of sexually transmitted diseases at Mulago National Referral Hospital in Uganda (ASTRHA): protocol for an open-label, randomised controlled trial. BMJ Open. 2024 Jun 11;14(6):e084806. doi: 10.1136/bmjopen-2024-084806. PMID 38862220